CLINICAL TRIAL: NCT02234557
Title: Movement-Based Training for Children With ADHD: A Feasibility Study
Brief Title: Tai Chi Training for Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21MH104651-01 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-09-09 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: ADHD
Keywords: Motor Control; Attention; Cognitive Control
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tai Chi (Experimental): Tai Chi instruction, 1 hour, twice per week Home Tai Chi practice with video, requesting 15-30 minutes, 3 times per week, monitored by practice log
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Tai Chi — 6-8 students will be enrolled in 8 weeks of Tai Chi instruction, with two 1-hour sessions per week. Students will be requested to practice from recorded materials at home three times a week for 15-30 minutes each session, and parents will be asked to keep a log of at-home practice.
  Class sessions will consist of warm up (qi k'ong), postural and breathing exercises, Tai Chi form practice, and Tai Chi games (including push hands).
  Practice will consist of warm up, followed by practice of selected pieces of the form.
  Children on stimulant medications will remain on these medications during the training period (though they will be asked to stop medications one day prior to motor and cognitive testing pre-, mid- and postintervention).
  Other Names: taichi; tai ji; taiji; t'ai chi; t'ai ji

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) has tremendous individual and societal impact, and the effectiveness of current standard treatments is limited. We examine a novel treatment that could remediate the core features of ADHD and thereby contribute to sustained improvements in behavioral control. This approach is motivated by mounting evidence that children with ADHD show difficulties with motor control, and that these motor deficits are strongly associated with the core behavioral features of ADHD. We employ Tai Chi, targeting improvements in well-established behavioral and physiologic measures of motor control, and with this, improvements in ADHD symptoms. The proposed study offers immense potential for the development of novel therapeutic approaches for ADHD with little risk of adverse reaction.

The over-arching goal of this proposal is to examine a movement-based mindfulness training as a therapeutic intervention for children with ADHD. This approach is motivated by two complimentary lines of evidence: 1) Children with ADHD show impairments in motor control that parallel (and correlate with) core deficits in behavioral control that define the disorder. 2) Gains in cognitive and behavioral control have been observed in adults learning Tai Chi, dance, or meditation. These lines of evidence provide substantial motivation for our proposed investigation of movement-based mindfulness training in children with ADHD. Specifically, we propose to evaluate an established Tai Chi-based intervention. We chose this approach for a number of reasons: 1) Tai Chi is among the most well-established movement-based interventions with documented therapeutic effects, including cognitive effects. 2) While many movement-based approaches show evidence of yielding cognitive improvements Tai Chi provides excellent opportunities for engagement of 8-12 year old children in the form of the collaborative game "push hands." 3) Tai Chi instruction consists of gentle movements that can be practiced even by those with physical limitations, and is readily available in the United States so the protocols developed in this study will be straightforward to deploy at a national level.

Hypothesis: After participating in a Tai Chi program, children with ADHD will show improvements in behavioral and physiologic measures of motor control. We further expect movement-based training will result in decreases in ADHD symptom severity.

DETAILED DESCRIPTION:
Persistent poor outcomes for individuals with ADHD make it imperative to explore intervention approaches beyond medication, particularly interventions that could provide sustained improvements in control of hyperactive, impulsive and distractible behavior. Two lines of evidence converge to support a movement-based mindfulness training intervention as a potential stand-alone or adjunct treatment for the treatment of ADHD symptoms. First, decades of research, including from our lab, has established that many children with ADHD show impairments in motor control that parallel their impairments in behavioral and cognitive control. Second, there is mounting evidence that movement-based mindfulness interventions are effective for enhancing behavioral control in adults, although there has been limited examination in children. These lines of evidence suggest an outstanding opportunity for development of novel treatment approaches for ADHD through engagement of the motor system.

In this application we propose to examine the efficacy of a specific movement-based mindfulness intervention for children with ADHD - Tai Chi. This approach was chosen for a number of reasons: 1) extensive documentation in the research literature, 2) engagement afforded by a martial approach to mindful movement, and 3) scalability given the existing availability of Tai Chi instruction in the United States and the ease of performing gentle Tai Chi movements even in the presence of physical limitation. Consistent with the "Fast-Fail" approach in the first two years (R21 phase) we will investigate the impact of Tai Chi on the motor system targets our lab has established as highly correlated with measures of classic ADHD symptoms. Specifically, we will measure SICI (short-interval intra-cortical inhibition via TMS) and overt movement behavior resulting from failures of motor control (mirror overflow and motor impersistence). Milestones will comprise successful motor system target engagement in the context of Tai Chi training. The findings will lay a foundation for the clinical exploration of Tai Chi and other movement-based mindfulness training approaches in ADHD and other conditions where the motor system is implicated. Our brain-based approach further provides a clear path for reliable assessment as well as integration with the cognitive neuroscience literature on inhibition and other aspects of cognitive control.

The motor system provides a locus for the integration of multiple neural systems, with clear abnormalities in inhibitory function in ADHD. An intervention targeting the motor system stands to make productive contact with these motor system targets. Indeed, there is broad evidence for the efficacy of Tai Chi (and other mindfulness-based movement training) in addressing a wide range of issues, including high level cognitive functions such as attentional control.2 The majority of these effects have been established in adults, but given the greater brain plasticity documented in children,1 we have reason to expect strong effects in children. Indeed, successes have been reported in child populations as early as preschool.32 Moreover, there is a recognized need for physiologic biomarkers in mindfulness and movement training studies.15 Our robust ability to track changes in specific motor markers at behavioral and physiologic (from TMS) levels, provides an ideal target measure to establish specificity in a Tai Chi training intervention.

Overview of intervention

Tai Chi is a form of exercise with a variety of components and a strong cultural tradition. In consultation with experienced teachers of Tai Chi, we have received consistent feedback that "martial applications," and specifically push hands, will likely be a valuable component of training for children with high distractibility. Central to the martial practice of Tai Chi is a collaborative game called "Push Hands," in which partners attempt to push one another off balance without the use of strong effort. Push hands, and other Tai Chi inspired "games" will be used to motivate engagement in slower, more focused movement training: Tai Chi warm-up, postural and breathing exercises, and a section of a Tai Chi form. We expect these components to collectively drive learning and development of behavioral control in the motor domain, with high potential for impact on other features of ADHD.

The Tai Chi instructor, a graduate student from the Johns Hopkins Tai Chi club, has extensive experience with youth instruction, as well as a keen understanding of the relationships between Tai Chi and "hard" martial arts from over 20 years of practice in martial arts, including 12 years of Tai Chi. An assistant instructor will additionally be engaged to assist with maintaining class focus. All instructors will be certified for ethical treatment of human subjects, as well as standards for youth physical education. Sessions will be held in an athletic facility on the Kennedy Krieger Institute (KKI) Greenspring campus. The athletic facility was designed and equipped for children with a range of abilities as part of the LEAP Program (Life-skills and Education for Students with Autism and other Pervasive Behavioral Challenges). It is advantageously located on a campus that is very convenient for most Baltimore area families. The facility moreover has a high-impact floating rubber floor. This environmentally friendly and slip-resistant flooring provides cushioning, which reduces fatigue and potential for injury to the participants during physical activities.

Recruitment and testing

Recruitment, preintervention data collection (see below for details), and logistical preparation will commence as early as is practicable once the funding period is established. At least three sessions will be completed, scheduled so as to ensure sessions both during the school year and during summer break. Six-eight students will be enrolled in each session, with a target of five-seven children successfully completing each session and participating in preintervention (three week period prior to the start of classes) , midpoint intervention (during weeks four-six of classes), and postintervention (the three weeks after classes complete) physiologic and behavioral assessments. Outcomes will be computed as the difference between preintervention and postintervention scores, while midpoint intervention scores will be used to give a sense of the timecourse of change for each measure.

It is expected that one student on average will be unable to successfully complete a given class series. Enrollment procedures will be adapted if necessary. As per our "intent to treat" approach (see below), children will be included in primary analyses irrespective of adherence to protocol (i.e., attendance). However, children may be requested to leave the class if their absence becomes disruptive. In total, we anticipate a minimum of 18 participants completing the training out of a total of 21 children enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Children must meet diagnostic criteria for ADHD on the Kiddie Schedule for Affective Disorders and Schizophrenia
* Comorbid oppositional defiant disorder (ODD) and simple phobias are permitted
* right handed
* Stimulant or no medication

Exclusion Criteria:

* left handed
* diagnosis of Intellectual Disability, Developmental Language Disorder, Reading Disability, or Autism (screened for using the Social Competence Questionnaire (SCQ)
* neurologic disorder (e.g., epilepsy, cerebral palsy, traumatic brain injury, Tourette Syndrome)
* documented hearing impairment ≥ 25 dB (decibel) loss in either ear.
* history of speech/language disorder or a Reading Disability (RD)
* a Full Scale IQ (Intelligence Quotient) score on the WISC-IV (Wechsler Intelligence Scale for Children) below 80
* a standard score below 85 on the Word Reading Subtest, regardless of IQ score
* foster care
* previous participation in Tai Chi Training
* parent and child report signs of puberty above Tanners-2
* Female participants will be excluded if they are pregnant or may be pregnant
* Non-stimulant psychoactive medications (e.g., atomoxetine, clonidine, tricyclic antidepressants, selective serotonin re-uptake inhibitors)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Motor persistence score | Change from baseline in total postintervention score, approx. 10 weeks
  A total score combining NEPSY ("A Developmental NEuroPSYchological Assessment") statue task and lateral gaze fixation.
  A halving of the distance from TD (Typically Developing) baseline for motor persistence measures (based on preexisting control data, and barring ceiling effects) will be regarded as a clinically meaningful change.

SECONDARY OUTCOMES:
TMS SICI (short-interval intracortical inhibition) | Change from baseline in total postintervention score, approx. 10 weeks
  SICI is obtained in paired pulse TMS trials, in which the first conditioning subthreshold pulse causes the subsequent suprathreshold pulse, on average, to evoke a smaller response in muscle. We expect this SICI effect to be diminished in ADHD preintervention (i.e., less of a reduction). Postintervention, we expect more robust SICI reduction in muscle response (i.e., more like the typically developing baseline).
  This will be compared to results from stimulant medication, in which patients recovered approximately half-way towards typically developing baseline.
Cognitive motor control | Change from baseline in total postintervention score, approx. 10 weeks
  RDoC (research domain criteria) battery for cognitive control targeting response inhibition delivered via laboratory computer (flanker task, Go / No-Go, and Stop Signal). We expect significant improvements across RDoC relevant scores.
Goniometer-based measures of sequential finger movements | Change from baseline in total postintervention score, approx. 10 weeks
  Mirror overflow, speed, and rhythmicity will be assessed with goniometers during simple sequential finger movements. We expect reductions in overflow postintervention. We will report on changes in other measures, but these are not central to our hypothesis.
Evaluation of Tai Chi performance | Change from baseline in total postintervention score, approx. 10 weeks
  Students will be asked to perform a subset of Tai Chi movements from the training, which will be scored on a 0-2 point scale for each movement. We expect performance to improve over the course of the intervention.

OTHER OUTCOMES:
Clinical measures of ADHD symptom severity and motor coordination | Change from baseline in total postintervention score, approx. 10 weeks
  We will administer Connors and DuPaul surveys (parent versions), the BASC-2 (Behavior Assessment System for Children, Second Edition, parent and child versions), and DCDQ (Developmental Coordination Disorder Questionnaire). We expect improvements on these measures over the course of the intervention. In particular, based on Hernandez-Reif, et al. (2001), we expect marked improvements on Connors subscales for Anxiety, Conduct, Daydream, Emotion, and Hyperactive.
Behavioral assessments of basic motor control | Change from baseline in total postintervention score, approx. 10 weeks
  We'll administer the PANESS (Physical and Neurologic Examination of Subtle Signs) and mABC-2 (Movement Assessment Battery for Children). We expect improvements over the course of the intervention.
Surveys of expectations | preintervention
  Prospective survey to assess expectations at outset. Results will be reported as descriptive statistics and representative text samples.
Surveys of Satisfaction | postintervention
  A retrospective survey to assess satisfaction and plans to continue with Tai Chi or other movement classes following the intervention. Results will be reported as descriptive statistics and representative text samples.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Mostofsky, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- LEAP Facility at Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Clark D, Seymour KE, Findling RL, Mostofsky SH. Subtle Motor Signs as a Biomarker for Mindful Movement Intervention in Children with Attention-Deficit/Hyperactivity Disorder. J Dev Behav Pediatr. 2020 Jun/Jul;41(5):349-358. doi: 10.1097/DBP.0000000000000795. PMID 32555070